CLINICAL TRIAL: NCT04814641
Title: Hypophosphatemia In Infants With Severe Bronchiolitis: Prevalence And Risk Factors
Brief Title: Hypophosphatemia and Bronchiolitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: A289
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Hypophosphatemia; Bronchiolitis
Keywords: Hypophosphatemia; Bronchiolitis; Paediatric Intensive Care Unit; Risk Factor
MeSH Terms: conditions — Hypophosphatemia; Bronchiolitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants with hypophosphatemia: Infant less than 3 months with severe bronchiolitis admitted in a pediatric intensive care unit, with hypophosphatemia in the first 5th days
  Interventions: Biological: hypophosphatemia occurrence in infants with severe bronchiolitis admitted in a pediatric intensive care unit
- Infants without hypophosphatemia: Infant less than 3 months with severe bronchiolitis admitted in a pediatric intensive care unit, without hypophosphatemia
  Interventions: Biological: hypophosphatemia occurrence in infants with severe bronchiolitis admitted in a pediatric intensive care unit

INTERVENTIONS:
Biological: hypophosphatemia occurrence in infants with severe bronchiolitis admitted in a pediatric intensive care unit — Serum phosphorus level < 1.55 mmol/L at any time between admission and the 5th day.

SUMMARY:
Bronchiolitis is a major public health problem and the leading cause of paediatric intensive care unit admission in infants. Hypophosphatemia is common in adult intensive care units and was associated with an increase of the duration of mechanical ventilation and the length of stay. Our hypothesis is that hypophosphatemia is common in bronchiolitis and could be a marker of severity.

ELIGIBILITY:
Inclusion Criteria:

* Age > 7 days and < 3 months of life
* Admission to the pediatric intensive care unit from 01/11/2016 to 31/03/2020
* With a diagnosis of moderate to severe bronchiolitis according to HAS 2019 criteria

Exclusion Criteria:

* Renal Failure and tubulopathy
* Previous disorder of phospho-calcium balance
* Malignant pathology
* Lenght of stay less than 24 hours
* History of cardiac, aortic or hepatic surgery

Ages: 7 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infant less than 3 months with severe bronchiolitis admitted in a pediatric intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-03-21 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
hypophosphatemia occurrence in severe bronchiolitis in infants admitted in a pediatric intensive care unit | At any time in the first 5th days after Pediatric intensive care admission
  A serum phosphorus level< 1.55mmol/L defines the hypophosphatemia.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Femme Mere Enfant - Groupement Hospitalier Est, Bron, France